CLINICAL TRIAL: NCT03976492
Title: The Research for New Clinical Diagnostic Strategy of Specific Biomarkers for Traumatic Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Baiyun Liu (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor-Investigator, Baiyun Liu, professor, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Other Study IDs: BTHospital KY2019-012-04
Record Dates: First submitted 2019-06-03; First posted 2019-06-06 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal group: normal population
- Brain injury group: patients with traumatic brain injury within 24 hours
  Interventions: Diagnostic Test: diagnostic of specific biomarkers
- Non-brain injury group: Non-brain injury group refers to patients with limb injury or systemic injury except brain injury.
  Interventions: Diagnostic Test: diagnostic of specific biomarkers

INTERVENTIONS:
Diagnostic Test: diagnostic of specific biomarkers — Protein and metabolic product differences will be detected from blood or lesion samples of normal population, patients with traumatic brain injury and/or non-brain injury using mass spectrometry proteomics and metabolomics analysis platform. Diagnostic markers of potential traumatic brain injury will be found, and their differential diagnostic values were discussed.
  Groups: Brain injury group; Non-brain injury group

SUMMARY:
Traumatic brain injury (TBI) is the most common type of nerve injury and it severely endangers the public health. It is necessary to accurately measure the early neurological function of brain injury for monitoring its prognosis and therapeutic interventions. Glasgow Coma Score (GCS) and Computed Tomography (CT) are often used to diagnose the severity of TBI. However, GCS has its drawbacks in the observation of prognosis, because it is interfered by analgesics, sedatives and relaxants in the evaluation of neurological function. CT may miss the diagnosis of diffuse axonal injury (DAI) and the monitoring of intracranial pressure (ICP). Secondary injuries after TBI, such as oxidative stress, inflammatory damage, and abnormal metabolism, can destroy cerebral blood vessels and structures, which also affect the diagnosis of injury. Therefore, there is an urgent need for new methods to quickly identify which patients are likely to suffer brain injury or even cause persistent disability. Detection of brain injury biomarkers based on blood and brain tissue has long been used to assess the severity of TBI, but no biomarkers have been found for early diagnosis of mTBI and prognosis of different degrees of brain injury. Protein and metabolic product differences were detected from blood or the lesion samples of normal population, patients with traumatic brain injury and/or non-brain injury using mass spectrometry proteomics and metabolomics analysis platform, and diagnostic markers of potential traumatic brain injury were found, and their differential and diagnostic values were discussed.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female, aged from 18 to 65.
2. Patients with brain injury within 24 hours after injury
3. Non-brain injury group refers to patients with limb injury or systemic injury except brain injury.
4. The subject reads and fully understands the instructions of the patients and signs the informed consent.

Exclusion Criteria:

1. Male or female, aged below 18.
2. Patients with definite history of central nervous system or cardiovascular system or taking drugs affecting the central nervous system.
3. Patients with severe metabolic diseases.
4. Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: normal population, patients with brain injury within 24h combined with or without systemtic injuries.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Protein levels of GFAP、UCH-L1、H-FABP、Aβ40、Aβ42、IL-10、NF-L、S100B and tau | One year
  The difference protein levels of GFAP、UCH-L1、H-FABP、Aβ40、Aβ42、IL-10、NF-L、S100B and tau assessed by the proteomics of the one year after traumatic brain injury.
Discovery of metabolic biomarkers in plasma that will lead to the early detection of traumatic brain injury | One year
  Metabolic biomarkers in plasma, such as methionine、glycine、cysteine、gamma-glutamylleucine、5-oxoproline、alpha-ketobutyrate、2-hydroxybutyrate, etal.. assessed by the metabolomics of the one year after traumatic brain injury.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
Published in the form of an article after the completion of the trail.